CLINICAL TRIAL: NCT00281411
Title: Follow-up Study of Endovascular Abdominal Aortic Aneurysm Treatment
Brief Title: Follow-up of Endovascular Aneurysm Treatment - The FEAT Trial
Status: Completed | Type: Observational
Sponsor: Clinical Research Office Imaging Division (Other)
Responsible Party: Sponsor-Investigator, Clinical Research Office Imaging Division, Clinical research coordinator, UMC Utrecht
Organization: UMC Utrecht (Other)
Other Study IDs: METC.2005.01.291E
Record Dates: First submitted 2006-01-20; First posted 2006-01-24 (Estimated); Last update posted 2018-02-15 (Actual); Status verified 2016-11

CONDITIONS: Aortic Aneurysm, Abdominal
Keywords: Blood Vessel Prosthesis Implantation; Endovascular aneurysm repair; Magnetic Resonance Angiography; Computed Tomography Angiography; Endoleak
MeSH Terms: conditions — Aortic Aneurysm, Abdominal; Endoleak

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Procedure: Computed Tomography Angiography — Computed Tomography Angiography
Procedure: Magnetic Resonance Angiography — Magnetic Resonance Angiography

SUMMARY:
After endovascular abdominal aortic aneurysm repair, life-long follow-up is needed to monitor the effectiveness of exclusion of the aneurysm sac from blood flow. For this reason, aneurysm diameter and the presence of endoleaks is evaluated with CT angiography yearly after Endovascular Aneurysm Repair (EVAR).

The aim of this study is to investigate the value of MRA examinations for the follow-up of these patients. The advantages of MRA with respect to CTA are no use of ionizing radiation, use of less nephrotoxic contrast agents.

DETAILED DESCRIPTION:
The FEAT trial (Follow-up of Endovascular Aneurysm Treatment) is designed as a prospective, single-center, follow-up study. 100 Patients will be enrolled in this study. These patients will undergo additional MRA-examinations the day before EVAR, the day after EVAR, 6 months and 1 year after EVAR. These patients also participate in the conventional CTA follow-up scheme which comprises a pre- and post-operative CTA and a CTA yearly thereafter. Coagulation parameters in the blood will be measured before and 1 year after EVAR.

ELIGIBILITY:
Inclusion Criteria:

* Patient is planned for endovascular abdominal aortic aneurysm repair

Exclusion Criteria:

* contraindication for MRI examination

  * claustrophobia
  * pacemaker
  * other non-MRI compatible implants

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient planned for endovascular abdominal aortic aneurysm repair
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2001-03; Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: W. Mali, MD PhD, Principal Investigator — UMC Utrecht
Locations (1):
- UMC Utrecht, Utrecht, Netherlands